CLINICAL TRIAL: NCT00894283
Title: A Pilot Study to Determine the Feasibility of Conducting a Randomized Clinical Trial Comparing Fondaparinux Sodium (Arixtra) Once Daily With Enoxaparin (Lovenox®) Twice Daily With Respect to Preventing VTE After Bariatric Surgery in Obese Patients
Brief Title: Comparing Enoxaparin to Fondaparinux to Prevent Venous Thromboembolism (VTE) in Bariatric Surgical Patients
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Prevention
Other Study IDs: NA_00025492
Record Dates: First submitted 2009-05-05; First posted 2009-05-06 (Estimated); Last update posted 2019-06-07 (Actual); Status verified 2019-06

CONDITIONS: Deep Venous Thrombosis; Pulmonary Embolism
Keywords: DVT; PE; MRV; bariatric surgery
MeSH Terms: conditions — Venous Thrombosis; Pulmonary Embolism | interventions — Enoxaparin; Fondaparinux

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Enoxaparin (Active Comparator): Patients will receive enoxaparin 40mg subcutaneously twice daily during perioperative period of bariatric surgery. Patients will be encouraged to ambulate and compression stockings while in bed.
  Interventions: Drug: Enoxaparin
- Fondaparinux (Active Comparator): Fondaparinux 5mg subcutaneously 6 hours following surgery, fondaparinux 5mg subcutaneously once daily during hospitalization. Patients will be encouraged to ambulate and compression stockings while in bed.
  Interventions: Drug: Fondaparinux

INTERVENTIONS:
Drug: Enoxaparin — Patients will receive enoxaparin 40mg subcutaneously twice daily during perioperative period of bariatric surgery. Patients will be encouraged to ambulate and compression stockings while in bed.
  Arms: Enoxaparin
Drug: Fondaparinux — Fondaparinux 5mg subcutaneously 6 hours following surgery, fondaparinux 5mg subcutaneously once daily during hospitalization. Patients will be encouraged to ambulate and compression stockings while in bed.
  Arms: Fondaparinux

SUMMARY:
This pilot study is designed to determine the feasibility of conducting a randomized clinical trial comparing fondaparinux sodium (Arixtra) once daily with enoxaparin (Lovenox®) twice daily with respect to preventing deep vein thrombosis (DVT) and pulmonary embolism (PE) after bariatric surgery in obese patients.

DETAILED DESCRIPTION:
In order to determine the feasibility of such a trial we need to determine the necessary sample size. In order to determine the necessary sample size, we need to obtain estimates of the incidence of DVT and the prevalence of PE using MRV in each treatment group. Descriptive statistics and 95% confidence intervals will be calculated to determine the incidence of DVT and the prevalence of PE using MRV in obese patients who have received treatment to prevent DVT and PE associated with bariatric surgery.

Anti-factor Xa levels will be used to help determine if treatments are reaching appropriate levels.

ELIGIBILITY:
Inclusion Criteria:

1. Men or women 18 years or older.
2. Body mass index (BMI) of 35kg/m2 or greater.
3. Undergoing laparoscopic bariatric surgery, i.e., laparoscopic sleeve gastrectomy, laparoscopic Roux-en Y gastric bypass or laparoscopic duodenal switch.

Exclusion Criteria:

1. History of previous deep vein thrombosis.
2. History of previous pulmonary emboli.
3. History of documented clotting/coagulation disorder.
4. History of cancer.
5. Weight < 50 kg or > 200 kg or unable to fit in MRI scanner.
6. Presence of metallic foreign bodies
7. Recent history of smoking (within the last year).
8. History of venous stasis disease.
9. History of obesity hypoventilation syndrome.
10. Patients who are unable to lay flat for extended periods of time or are claustrophobic.
11. Patients who have a pacemaker, an implanted defibrillator or certain other implanted or electronic or metallic devices (implanted medical or metallic devices, shrapnel, or metal).
12. History of hypersensitivity reaction to anticoagulation products.
13. History of HIT (Heparin Induced Thrombocytopenia.
14. History of Renal Insufficiency (Creatinine Clearance < 50).
15. Active clinically significant bleeding.
16. Acute bacterial endocarditis.
17. BMI > 60.
18. Patients with metallic foreign body or implant (unable to have an MRV study).

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2009-06; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
To estimate the prevalence of asymptomatic deep venous thrombosis and pulmonary emboli in obese patients undergoing bariatric surgery. | 2 years

SECONDARY OUTCOMES:
To assess the relationship of Anti-factor Xa levels and the occurrence of deep venous thrombosis and pulmonary emboli in bariatric patients receiving standard dose of anticoagulation (enoxaparin/Lovenox or fondaparinux/Arixtra). | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kimberley E Steele, MD, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Bayview Medical Center, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Amaral FC, Baptista-Silva JC, Nakano LC, Flumignan RL. Pharmacological interventions for preventing venous thromboembolism in people undergoing bariatric surgery. Cochrane Database Syst Rev. 2022 Nov 22;11(11):CD013683. doi: 10.1002/14651858.CD013683.pub2. PMID 36413425